CLINICAL TRIAL: NCT05643183
Title: Innovative Healthcare Delivery for Patients With Asthma by Means of Digitally Supported Self-management: A Pilot Study in Secondary Care
Brief Title: Digitally Supported Self-management Program for Patients With Asthma in Secondary Care: a Pilot Study
Acronym: Astmakompas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, jjaardoom, Dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL80559.058.22; 10390052010011 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Asthma
Keywords: Asthma control; Uncontrolled asthma; Asthma; Self-management; Application; eHealth; mHealth
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving Astmakompas (Experimental): 30 patients from two hospital sites (AMC and MST)
  Interventions: Other: Astmakompas

INTERVENTIONS:
Other: Astmakompas — The Astmakompas platform consists of a patient app, a portal for HCPs, and a wireless spirometer connected to the patient app. The patient app combines monitoring with self-management tools, and provides a portal to present these data as well as to communicate with their HCP. Patients' monitoring data is linked to their personalized digital action plan, including self-management strategies and treatment recommendations based on the latest international treatment guidelines. The action plan aims to increase patients' awareness of their symptoms and/or the severity of their symptoms, as well as their corresponding adverse effects. When patients' monitoring results show a deterioration of asthma control, HCPs receive smart notifications. Patient data can thereby serve as direct input in the consultations with the HCP, or they can proactively offer as-needed support. Patients are able to ask non-critical asthma-related questions to their HCP through a chat function of the application.

SUMMARY:
In the Netherlands, more than 600 thousand people have asthma. About half of these people have insufficient asthma control. This has a negative effect on their health and use of care. Insufficient knowledge about asthma and proper medication use, low self-confidence in managing asthma, and low compliance contribute to this problem. AstmaKompas is an eHealth application for asthma patients focused on self-monitoring and self-management. Astmakompas also connects patients with their healthcare professionals, among other things by giving healthcare professionals more insight into their patients' disease progression, enabling them to provide timely(er) support. In this study, AstmaKompas will be deployed and evaluated in 2 hospitals. Through questionnaires and interviews, insight will be gained into the experiences of patients and healthcare professionals with AstmaKompas. Potential effects on health outcomes and healthcare utilization will also be identified.

DETAILED DESCRIPTION:
Asthma is a major chronic disease that is estimated to affect approximately 262 million people worldwide. Asthma control is often suboptimal, with approximately 50% of patients having (partially) uncontrolled asthma. These patients have a higher risk of asthma exacerbations, asthma-related hospitalization and emergency department visits, resulting in high healthcare and societal costs. Poor asthma control is furthermore a major contributor to impaired health-related quality of life. Although the literature shows promising results of (digital) supported self-management interventions in improving asthma control and other important health outcomes, relatively little is known about the cost-effectiveness of such supported digital interventions delivered on a smartphone in comparison to usual care. Furthermore, no cost-effectiveness research has been conducted in a secondary care.

The primary aim of the proposed pilot study is to investigate whether Astmakompas is feasible, acceptable, easy and safe to use in a secondary care context for both patients and healthcare professionals (HCPs). The secondary aim is to explore the potential effect of Astmakompas on health and healthcare outcomes. Study design: A mixed-method study consisting of a multi-center, single-arm, pre-post intervention study with a duration of 12 weeks. The quantitative part consists of a survey providing insights on the feasibility, acceptability, usability, safety, and preliminary effects of Astmakompas. The explanatory qualitative part consist of semi structured focus groups for patients, and individual interviews for HCPs, which will complement the quantitative results.

The researchers aim to recruit a total of 30 patients in two hospitals: 15 in the Amsterdam UMC location AMC, and 15 in Medisch Spectrum Twente (MST). Inclusion criteria are 1) being aged 18 years or older, 2) not having used Astmakompas before, 3) having a physician diagnosis of asthma, 4) having uncontrolled asthma as defined by a score of 1.5 or higher on the Asthma Control Questionnaire (ACQ), 5) being able to understand, read and speak the Dutch language (i.e., based on self-report), and 6) having access to the Internet and a smartphone. Exclusion criteria are having a respiratory disease other than asthma, or having a non-reversible airway obstruction. Four involved HCPs (i.e., one pulmonologist and one pulmonary nurse in each of the two participating hospitals) will be invited to participate in the interviews.

Astmakompas is a CE-certified eHealth application for patients with asthma. The platform consists of a patient app, a portal for HCPs, and a wireless spirometer connected to the patient app. The patient app combines monitoring with self-management tools, and provides a portal to present these data as well as to communicate with their HCP. The monitoring enables patients to monitor their asthma control on a weekly basis using a standardized Patient Reported Outcome Measure (PROM) questionnaire, and additionally with a spirometer that assesses, amongst others, FEV1 and FVC. Patients' monitoring data is linked to their personalized digital action plan, including self-management strategies and treatment recommendations based on the latest international treatment guidelines. The action plan aims to increase patients' awareness of their symptoms and/or the severity of their symptoms, as well as their corresponding adverse effects. The action plan subsequently supports patients to intervene in a more timely manner, thereby preventing worsening of symptoms. When patients' monitoring results show a deterioration of asthma control, HCPs receive smart notifications by means of algorithms. Patient data can thereby serve as direct input in the consultations with the HCP, or they can proactively offer as-needed support. Patients are able to ask non-critical asthma-related questions to their HCP through a chat function of the application.

Primary study parameters include the Feasibility of Intervention Measure (FIM), the Acceptability of Intervention Measure (AIM, only administered to HCPs), user patterns of Astmakompas (e.g., number of logins), the Client Satisfaction Questionnaire-8 (CSQ-8, only administered to patients), the System Usability Scale (SUS, administered to both HCPs and patients), and adverse events (assessed in patients). Qualitative assessment in patients and HCPs will give a more in-depth understanding of feasibility, acceptability, usability and safety. Secondary study parameters, all assessed in patients, include asthma control (assessed using the Asthma Control Questionnaire [ACQ] and the weekly monitoring questionnaire that is part of Astmakompas), lung function as assessed by the spirometer, the Respiratory Illness questionnaire-Monitoring 10 (RIQ-MON10), the EuroQol 5 dimensions 5 levels (EQ-5D-5L), the Perceived Control of Asthma Questionnaire (PCAQ), and items from the iMTA Productivity Cost Questionnaire (iPCQ) and iMTA Medical Consumption Questionnaire (iMCQ). Additionally, qualitative assessment in patients and HCPs will give a more in-depth understanding of direct and indirect costs.

Regarding time investment, all participating asthma patients will be asked to complete a questionnaire at baseline, taking approximately 15-20 minutes, and at post-intervention (i.e., 12 weeks after baseline), taking approximately 25 minutes. Furthermore, part of the Astmakompas intervention is completing a weekly questionnaire taking approximately 2-3 minutes to complete, and weekly spirometer assessments (i.e., approximately 1-5 minutes each). In addition, a subsample of patients (n = 8 to 12) will participate in an online focus group interview lasting approximately 90 minutes, which will be reimbursed with a gift voucher of 25 euro. In line with the experiences of two previous small pilot studies, the researchers do not expect any health risks to be associated with the use of Astmakompas. Potential benefits include increased asthma control and self-management of the disease, as well as more efficient care by means of among others increased access to medical staff. Hence, the potential benefits are expected to outweigh the burden of the study. The participating four HCPs will participate in an individual interview lasting 60 minutes, which will be reimbursed with a gift voucher of 100 euro

ELIGIBILITY:
Inclusion Criteria:

Being aged 18 years or older Not having used Astmakompas before Having a physician diagnosis of asthma Having uncontrolled asthma as defined by a score of ≥ 1.5 on the ACQ [19] Being able to understand, read and speak the Dutch language (i.e., based on self-report) Having access to the Internet and a smartphone

Exclusion Criteria:

Having a respiratory disease other than asthma Having a non-reversible airway obstruction

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of Astmakompas according to patients and HCPs. | After 12 weeks
  Feasibility of the intervention at post-intervention according to patients and HCPs.
Acceptability of Astmakompas according to patients and HCPs. | After 12 weeks
  Acceptability of the intervention according to HCPs will be assessed at post-intervention using the 4-item Acceptability of Intervention Measure (i.e., AIM). Patients' satisfaction with Astmakompas at post-intervention will be assessed using the 8-item Client Satisfaction Questionnaire (CSQ-8).
Usability of Astmakompas according to patients and HCPs. | After 12 weeks
  User-friendliness of Astmakompas will be assessed at post-intervention. In patients, the System Usability Scale (SUS) will be used to determine the user-friendliness of the Astmakompas intervention. In HCPs, the SUS will be used to determine the user-friendliness of the Astmakompas healthcare portal.
Safety of Astmakompas according to patients and HCPs. | After 12 weeks
  At post-intervention, an open-ended question will assess whether patients have experienced any negative effects due to their participation in Astmakompas.

SECONDARY OUTCOMES:
Asthma control in patients | First day and after 12 weeks
  The 6-item ACQ is used to assess asthma control in patients at baseline and post-intervention.
Rescue medication use in patients | First day and after 12 weeks
  The use of rescue medication usage during the intervention period will be assessed by an item in the monitoring questionnaire of Astmakompas.
(Asthma related) Quality of Life (QoL) in patients | First day and after 12 weeks
  The Respiratory Illness Questionnaire-Monitoring 10 will be used to assess asthma-related QoL at baseline and post-intervention. QoL will be measured with the EuroQol 5 dimensions 5 levels (EQ-5D-5L) at baseline and post-intervention.
Self-efficacy regarding perceived ability to manage and control asthma in patients | First day and after 12 weeks
  The 6-item version of the Perceived Control of Asthma Questionnaire (PCAQ) will be used to assess individuals' perceived confidence in their ability to manage their asthma and exacerbations effectively. The questionnaire consist of six items rated on a 5-point Likert scale. The total PCAQ-score is the sum score of the six items (total score range 6 - 30), whereby negatively worded items will be reverse scored so that higher scores represent greater perceived ability and confidence to manage and control asthma. Self-efficacy will also be discussed in focus-groups.
(In)direct costs by/in patients | First day and after 12 weeks
  Several items from the iMTA Productivity Cost (iPCQ) questionnaire will be administered at baseline and post-intervention to assess the impact of disease on absence from work in the past three months. Furthermore, several items of the iMTA Medical Consumption Questionnaire (iMCQ) will be used to assess patients' asthma-related healthcare consumption in the past three months, among others the number of visits to the general practitioner and hospital due to their asthma. (In)direct costs will also be discussed in focus-groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jiska Aardoom, Dr., Principal Investigator — Leiden University Medical Center (LUMC)
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No